CLINICAL TRIAL: NCT06884709
Title: Activity-based Mirror Therapy for Lower Limb Motor Recovery, Balance, Gait, and Mobility in Acute Inpatient Stroke: A Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 348947
Record Dates: First submitted 2025-02-24; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: stroke; acute stroke; mirror therapy; lower limb hemiparesis; stroke rehabilitation; stroke physiotherapy
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mirror Therapy Group (Experimental): For 15 minutes, three days per week for two weeks, participants will complete activity-based exercises with their non-paretic lower limb whilst watching the reflection of this limb in a mirror that is placed in their mid-sagittal plane.
  They will also receive 45 to 60 minutes of usual personalized conventional physiotherapy five days per week.
  Interventions: Other: Mirror Therapy

INTERVENTIONS:
Other: Mirror Therapy — During mirror therapy, participants will sit in an arm chair with a mirror placed in their mid-sagittal plane so that their non-paretic lower limb is reflected and their paretic lower limb is hidden. They will be asked to complete activity-based exercises with their non-paretic limb whilst watching the reflection in the mirror and imagining the reflection is their paretic limb.
  The activity-based exercises consist of rocker board dorsi/plantarflexion, rocker board in/eversion, step ups, wiping floor (or ball rolling) in/external hip rotation, wiping floor ab/adduction, ball kicking, and picking up marbles with the toes. Participants will do these exercises for 15 minutes, three days per week for four weeks.
  Participants will also receive 45 to 60 minutes of usual personalized conventional physiotherapy such as neurodevelopmental facilitation, sensory motor re-education, active/active-assisted exercises, and balance/gait training, five days per week.

SUMMARY:
This feasibility study is the first step of a larger effects study exploring the use of an activity-based mirror therapy program for people who have had a stroke in the last 30 days and are in the hospital. The study aims to examine features of the study design as well as the preliminary effects of the mirror therapy program on motor recovery, balance, gait, and mobility.

In this study participants will complete 15 minutes of lower limb mirror therapy three days per week for two weeks, alongside their usual physiotherapy. The motor recovery, balance, gait, and mobility of participants will then be reassessed. Participants will also be invited to complete a short questionnaire and interview about their experience in the study.

Stroke physiotherapists that are involved in the study will also complete a questionnaire and interview to provide feedback on the study and it's design.

DETAILED DESCRIPTION:
This study will recruit participants that are inpatients at the Queen Elizabeth University Hospital in Glasgow. Participants will be screened according to eligibility criteria. For example, participants must be between 72 hours and 30 days post-stroke at the time of baseline assessment and have hemiparesis or hemiplegia of the lower limb.

After providing written informed consent, participants will receive activity-based mirror therapy for 15 minutes, three days per week for two weeks, in addition to 45 to 60 minutes of usual personalized conventional physiotherapy five days per week. The mirror therapy will be conducted by Glasgow Caledonian University (GCU) Doctorate of Physiotherapy (DPT) student Cassidy Flammang under the supervision of a qualified physiotherapist, while the conventional physiotherapy will be conducted by the qualified physiotherapists on the stroke rehabilitation ward.

The mirror therapy sessions will involve the participants sitting in a chair with a back, arm rests, and optional side supports, with their hips, knees, and ankles positioned at 90°. A 60 cm X 165 cm mirror will be placed in the midsagittal plane so that the non-paretic limb is reflected. The participants will be instructed to view the reflection in the mirror whilst conducting activity-based exercises with the non-paretic limb. They will be further instructed to imagine that the reflection of the non-paretic limb is their paretic limb, but to keep their paretic limb still. The exercises will target all major lower limb movements, except hip extension as that cannot be addressed whilst seated. The exercises will consist of 10-15 repetitions each of the following: rocker board dorsi/plantarflexion, rocker board in/eversion, step ups, wiping floor (or ball rolling) in/external hip rotation, wiping floor ab/adduction, ball kicking, and picking up marbles with the toes. Participants may take up to one minute of rest between exercises. Participants will be informed that they can take breaks or skip exercises at any point.

Lower limb motor recovery, balance, gait, and mobility will be assessed at baseline and upon completion of the two-week intervention. Mean differences will be determined to assess the change in test scores from pre- to post-intervention using a paired t-test, if normally distributed, or a Wilcoxon sign rank test if not. Both would have a significance level of p<0.5.

Participants and physiotherapists involved in the study will also be asked to complete a short questionnaire and semi-structured interview to discuss the study and mirror therapy program. The interviews will be audio-recorded, with consent, and conducted by GCU DPT student Cassidy Flammang. They will then be transcribed and analyzed by thematic content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosis of hemorrhagic or ischemic stroke by head computed tomography (CT) or magnetic resonance imaging (MRI)
* Medically stable to participate in physical rehabilitation as determined by the medical staff at QEUHSRU providing approval to begin physiotherapy
* Between 72 hours and 30 days post stroke at the time of baseline assessment
* Hemiparesis or hemiplegia of lower limb
* Ability to maintain sitting balance in a chair with arm rests, a back, and optional side support while moving the lower limb
* Ability to ambulate with or without a walking aide prior to stroke
* No cognitive impairment that affects the ability to interact with the intervention or provide informed consent, as determined by the potential participant's medical team. To further ensure participants remain cognitively capable throughout the study, participants will be asked to briefly explain the study before providing consent and before each mirror therapy session
* No severe aphasia that would impair the participants ability to understand the instructions of the intervention or prevent them from providing continuous verbal feedback throughout the intervention. This will be determined by the potential participant's care team. To further ensure potential participants are not aphasic they will be asked to briefly being able to explain the study back to the research team prior to providing written consent and before each mirror therapy session
* No severe uncorrected visual impairments that would prevent viewing the image in the mirror
* No severe cardiopulmonary or musculoskeletal impairments that inhibit seated exercises of the non-paretic limb

Exclusion Criteria:

* Individuals with any type of lower limb amputation of either side of the body
* Individuals who have been identified as having incapacity by their medical team, as aligned with the Adults with Incapacity (Scotland) Act 2000
* Non-English Speakers
* Individuals who's care teams identified them as being distressed during their routine assessments/sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-04 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment Rate | Baseline
  Average monthly recruitment rate (total number of people approached about the study ÷ the number of months recruitment was conducted)
Participant Enrolment Rate | Baseline
  Average monthly enrolment rate (number of patient participants that provided written consent ÷ the number of months recruitment was conducted)
Rate of Recruitment to Enrolment | Baseline
  Recruitment to enrolment success rate (number of patient participants enrolled ÷ number of patient participants approached)
Participant Retention Rate | From baseline to the end of the intervention at 2 weeks
  Retention Rate (number of participants that completed the entire two-week intervention ÷ number of enrolled participants)
Participant Drop-out Rate | From baseline to the end of the intervention at 2 weeks
  Drop-out rate (number of participants that did not complete the entire two-week intervention ÷ number of enrolled participants)
  The number of participants that did not complete the entire two-week intervention will then by further broken down and analyzed for the following categories:
  * Dropped out of study on own volition
  * Withdrawn from the study due to medical complications, cognition/aphasia regression, or death
  * Discharged from the stroke ward during the two-week intervention
Outcome Measure Practicality: Outcome Measure Completion Rate (Pre-intervention) | Baseline
  Pre-intervention outcome measure completion rate (number of times each effects outcome measure was fully completed at baseline ÷ number of times each effects outcome measure was attempted at baseline)
Outcome Measure Practicality: Outcome Measure Completion Rate (Post-Intervention) | End of the intervention at 2 weeks
  Post-intervention outcome measure completion rate (number of times each effects outcome measure was fully completed post-intervention ÷ number of times each effects outcome measure was attempted post-intervention)
Data Collection Method Practicality: Conventional Physiotherapy Spreadsheet Completion rate | End of the intervention at 2 weeks
  Conventional physiotherapy spreadsheet completion rate (number of times the spreadsheet was successfully and fully filled out ÷ total number of sessions completed)
Data Collection Method Practicality: Mirror Therapy Tolerability Form Completion rate | End of the intervention at 2 weeks
  Mirror therapy tolerability form completion rate (number of times the form was successfully and fully filled out ÷ total number of sessions completed)
Data Collection Method Practicality: Physiotherapist Interview | Through study completion, up to 22 weeks
  Semi-structured interviews with the physiotherapists involved in the study to discuss the practicality of the data collection methods used in the study
Participant Acceptability of the Intervention: Participant Questionnaire | End of the Intervention at 2 weeks
  Participant acceptability questionnaire to assess how acceptable participants found the intervention. The questionnaire was adapted from Sekhon, Cartwright, and Francis' 2022 theoretical framework of acceptability informed questionnaire for healthcare interventions.
Participant Acceptability of the Intervention: Participant Interview | End of the Intervention at 2 weeks
  Semi-structured interviews with participants to discuss how acceptable participants found the intervention.
Physiotherapist Acceptability of Study: Physiotherapist Questionnaire | Through study completion, up to 22 months
  Physiotherapist acceptability questionnaire to assess how acceptable the stroke physiotherapists found the study and it's design. The questionnaire was adapted from Sekhon, Cartwright, and Francis' 2022 theoretical framework of acceptability informed questionnaire for healthcare interventions.
Physiotherapist Acceptability of Study: Physiotherapist Interviews | Through study completion, up to 22 months
  Semi-structured interviews with the physiotherapists involved in the study to assess how acceptable they found the study and it's design
Intervention Tolerability: Completion Rate of Each Mirror Therapy Exercise | End of the intervention at 2 weeks
  Completion rate of each mirror therapy exercise (number of times each individual mirror therapy exercise was completed in full ÷ total number of mirror therapy sessions)
Intervention Tolerability: Completion Rate of Entire Mirror Therapy Session | End of the intervention at 2 weeks
  Completion rate of entire 15-minute mirror therapy session (number of times the entire mirror therapy was completed in full (no skipped exercises) ÷ total number of mirror therapy sessions)
Intervention Tolerability: Participant Interviews | The end of the intervention at 2 weeks
  Semi-structured interviews with participants to discuss how tolerable they found the intervention.
Intervention Practicality: Average Weekly Amount of Conventional Physiotherapy Recieved | End of Intervention at 2 weeks
  Average amount of conventional physiotherapy participants recieved per week (in minutes)
Intervention Practicality: Average Weekly Amount of Mirror Therapy Recieved | End of Intervention at 2 weeks
  Average amount of Mirror Therapy participants recieved per week (in minutes)
Intervention Practicality: Physiotherapist Interview | Through study completion, up to 22 months
  Semi-structured interviews with stroke physiotherapists involved in the study to discuss the practicality of implementing the intervention with the given dosage and design.
Adverse Events | From baseline to the end of the intervention at 2 weeks
  What is it assessing?
  * Assesses if the participants experienced any adverse events throughout the study How is it Measured?
  * Participants will be asked about adverse events (related or unrelated to the intervention) at the beginning and end of each mirror therapy session. This will be recorded on the mirror therapy tolerability form.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment - Lower Extremity (FMA-LE) | Baseline and the end of the intervention at 2 weeks
  Assesses lower limb motor recovery. There is a maximum score of 34. A higher scores indicates better motor recovery.
Berg Balance Scale (BBS) | Baseline and the end of the intervention at 2 weeks
  Assesses balance. It consists of 14 items on a five-point ordinal scale that ranges from 0 to 4. 0 represents the lowest level of function and 4 the highest. There is a maximum score of 56.
10-Meter-Walk-Test (10MWT) | Baseline and the end of the intervention at 2 weeks
  Assesses gait. A 10 meter (m) walkway will have a 2 m acceleration and deceleration zone on each side. Thus the time (in seconds) taken to walk the central 6 meters will be measured, with speed calculated in m/s. This study will complete 1 trial at a comfortable speed
Modified Rivermead Mobility Index (MRMI) | Baseline and the end of the intervention at 2 weeks
  Assesses mobility. The MRMI assesses 8 mobility activities on a six-point scale from 0 to 5, with 0 being unable and 5 independent. There is a maximum score of 40. This study will assess some of the activities concurrently with the BBS and 10MWT.

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Joshi, PhD, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers. It will be stored on a password protected OneDrive that only the researchers of this study will have access to.